CLINICAL TRIAL: NCT00605449
Title: Phase I, Randomized, Open-Label, 3 Period Crossover Drug Interaction Study Between Simvastatin and GSK376501 in Healthy Subjects
Brief Title: A Drug Interaction Study Between Simvastatin and GSK376501
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DIX109980
Record Dates: First submitted 2008-01-18; First posted 2008-01-31 (Estimated); Last update posted 2010-10-19 (Estimated); Status verified 2010-10

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: GSK376501; Simvastatin; Healthy Subjects; Repeat Dose; Drug Interaction; Randomized; Pharmacokinetics
MeSH Terms: conditions — Diabetes Mellitus, Type 2

INTERVENTIONS:
Drug: GSK376501

SUMMARY:
This study is a 3-period crossover drug interaction study between GSK376501 and simvastatin in healthy adult subjects. This study will examine if repeat doses of GSK376501 affects the pharmacokinetics of simvastatin and if repeat doses of simvastatin affects the pharmacokinetics of GSK375601.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a responsible physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator considers that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Male or female between 18 and 55 years of age.
* A female subject is eligible to participate if she is of non-childbearing potential, defined as:

  * pre-menopausal females with a documented tubal ligation or hysterectomy; or
  * postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 MlU/ml and estradiol < 40 pg/ml (<140 pmol/L) is confirmatory].
* Body weight ≥ 50 kg and BMI within the range 19 - 30 kg/m2 (inclusive).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Demonstrates an average QTc interval < 450 msec (or < 480 msec in subjects with Bundle Branch Block), an average PR interval < 200 msec, and a QRS duration < 110msec (manual or machine read) at screening or baseline

Exclusion Criteria:

* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* A positive test for HIV antibody.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Previous exposure to GSK376501.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subjects will be excluded if they experience symptomatic or asymptomatic arrhythmia of any clinical significance during screening.
* The subject has a positive pre-study drug/alcohol screen and is unwilling to abstain from 72 hours prior to dose until follow-up. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines.
* Urinary cotinine levels indicative of smoking or history or use of tobacco or nicotine-containing products within 6 months prior to screening.
* Has a history of alcohol abuse or dependence within 12 months prior to the study. Alcohol abuse is defined as an average consumption of greater than 7 drinks per week for women or greater than 14 drinks per week for men. One alcohol drink is defined as the equivalent of 12 g of alcohol as follows: 5 oz/150 ml wine, 12 oz (360 ml) beer or 1.5 oz (45 ml) of 80 proof distilled spirits.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort, kava, ephedra [ma huang], gingko biloba, DHEA, vohimbe, saw palmetto, ginseng, red yeast rice) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication and is unwilling to abstain from use of these medications until the last pharmacokinetic sample has been collected, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* Use of caffeine- or xanthine-containing products for 24 hours prior to the start of dosing until collection of the final pharmacokinetic and sample of each study period.
* Consumption of any food or any beverage containing alcohol, grapefruit or grapefruit juice, apple or orange juice, Seville oranges, vegetables from the mustard green family (e.g., kale, broccoli, watercress, collard greens, kohlrabi, brussels sprouts, mustard) and charbroiled meats from 7 days prior to the first dose of study medication until the last pharmacokinetic sample has been collected.
* Use of acetaminophen within 48 hours of the first dose and is unable or unwilling to discontinue use of acetaminophen until the last pharmacokinetic sample has been collected.
* Use of aspirin, aspirin-containing compounds, salicylates or nonsteroidal anti-inflammatory drugs (NSAIDs) within 48 hours days of the first dose and is unwilling to abstain from use of these medications until the last pharmacokinetic sample has been collected.
* Use of liquid antacids (e.g. Maalox, Mylanta, Amphogel, milk of magnesia) or chewable antacids (e.g. TUMS) within 48 hours of the first dose and is unwilling to abstain from use of these medications until the last dose of study medication.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Alkaline phosphatase value higher than 1.5 times the upper limit of normal at screening or at baseline.
* Aspartate aminotransferase (AST), alanine aminotransferase (ALT), direct (conjugated) bilirubin, or CPK values higher than 1.25 times upper limit of normal at screening or at baseline.
* Fasting triglyceride level > 400 mg/dL (4.52 mmol/L) at screening or at baseline.
* Donation of blood or blood products in excess of 500 mL within a 56 day period.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* History of rhabdomylosis.
* History of or current congestive heart failure (NYHA Class I-IV symptoms - refer to Appendix 3)
* History of thyroid dysfunction or an abnormal thyroid function test as assessed by TSH as screening.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2008-01; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
drug plasma levels of GSK376501: | Day 7 Periods 1, 2 & 3

SECONDARY OUTCOMES:
drug plasma levels of GSK376501: | Day 7 all periods
adverse events, vital signs, con meds: | each visit, all periods
labs: | Days 4 & 8 all periods
ECGs: | Days 1-7 all periods
Simvastatin acid Day 7 tmax and t1/2.
Simvastatin Day 7 AUC(0-24), Cmax, tmax and t1/2.
GSK376501 Day 7 AUC(0-24), Cmax, tmax and t1/2.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, MPH, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Austin, Texas, United States